CLINICAL TRIAL: NCT04434495
Title: Outcome of Platelet Rich Plasma Injection in ICSI Patients, a Randomized Controlled Trial
Brief Title: Outcome of Platelet Rich Plasma in ICSI Patients, a Randomized Controlled Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Osman Hospital (Other)
Responsible Party: Principal Investigator, Dr Hisham Gouda, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DrOsmanH
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy Outcome
Keywords: PRP, IVF

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental): mock embryo transfer and PRP injection
  Interventions: Biological: PRP
- control group (No Intervention): only mock embryo transfer

INTERVENTIONS:
Biological: PRP — PRP injection into uterine cavity
  Arms: PRP group

SUMMARY:
2 groups randomized to PRP injectioninto uterine cavity at mock embryo transfer, and a control group with only mock embryo transfer.

DETAILED DESCRIPTION:
Participants are allocated in two groups ( randomized). Study is conducted in Dar El Teb infertility and IVF centre, Egypt. Normoresponder patients (9-15 mature follicles on day of HCG administration) and candidates for fresh embryo transfer are recruited to the study. 788 patients will be randomized on the day of ovum pick up in a 1 to 1 ratio to platelet rich plasma (PRP) group and control group. Patients wee randomized using computer generated randomization list and sequentially numbered sealed envelopes containing allocation information written on a card. The embryologist and doctors responsible for follow up after ovum pick up aew blinded to received treatment. Ovarian stimunlation is achieved by highly purified urinary FSH (Fostimon, IBSA, Switzerland)started on the 2nd or 3rd day of menstruation. The initial dose ranged between 150-300IU/d depending on expected ovarian response and serum E2 level. GnRH antagonist (Cetrotide, Serono international, Geneva, Switzerland) 0.25mgSC/day will be give when the leading follicle is 14mm and continued till day of HCG. 10,000 IU HCG will be given when 3 or more follicles are 18mm on mean diameter. Oocyte retrieval will be performed 34-36 hours after HCG administration. In PRP group, 1 ml autologous PRP prepared from blood of participants and injected under ultrasound guidance inside the uterus while performing the mock embryo transfer. In control group, mock embryo transfer was performed without injecting anything inside the uterus. All participants will receive progesterone vaginal pessaries (Prontogest, Marcyrl, Egypt) 400 mg twicw daily, starting on day of oocyte retrieval till 12weeks gestation or negative pregnancy test. No more than 3 embryos will be transferred2-5 days after oocyte retrival. B HCG levels will be measured in blood 14 days after HCGadministration. Transvaginal ultrasound will be performed 4 weeks after embryo transfer to confirm clinical pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Normoresponder patients (i.e. patients with 9 to 15 mature follicles on the day of HCG administration ) with expected good reproductive outcomes of IVF-ET and candidates for fresh embryo transfer

Exclusion Criteria:

* Age less than 18 years and more than 35 years Body mass index more than 30kg/m2 Serum progesterone level less than 1.5 ng/ml on the trigger day Smoking Moreover, patients with previous IVF cycle, PCOS ( polycystic ovarian syndrome), pelvic inflammatory disease, endometriosis, uterine anomalies, Ashermann syndrome, chronic endometritis, chromosomal anomalies, increased peripheral NK cells, hereditary thrombophylia and antiphospholipid syndrome were excluded from the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 788 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2020-11-15 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Four weeks post intervention
  The presence of gestational sac by transvaginal ultrasound

SECONDARY OUTCOMES:
Implantation rate | Four weeks post intervention
  The number of gestational sacs detected by ultrasound divided by the number of embryos transferred
Ongoing pregnancy rate | Five months post intervention
  Number of continued pregnancies beyond 20 weeks gestation
Abortion rate | Five months post intervention
  Number of pregnancies terminated before 20 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Gouda, MD, Principal Investigator — Assistant prof Cairo university

IPD SHARING:
Plan to Share IPD: No